CLINICAL TRIAL: NCT04446156
Title: Epidemiological Investigation of HIV-infected Patients Complicated With Liver Disease in Zhejiang Province
Brief Title: Liver Diseases in PLWH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: ZJHIVER
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: HIV/AIDS; Liver Diseases
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Liver Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In Highly Active Antiretroviral Therapy era, fatty liver has become an important cause of liver function damage in people living with HIV (PLWH). There are a large number of PLWH in China who are infected with hepatitis B virus and hepatitis C virus. HIV, hepatitis B virus, hepatitis C virus, drugs, alcohol, etc. affect each other, which makes the cause, diagnosis, and treatment of liver function damage in PLWH complicated in China.

The investigators plan to conduct a large-scale questionnaire survey among PLWH in Zhejiang Province to assess liver function, detect liver Injuries early, and analyze HIV, hepatitis B virus, hepatitis C virus, anti-HIV drugs, alcohol and other factors associate with liver injuries in PLWH, to provide basis for the treatment and prevention of liver disease in PLWH in eastern China.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* Non-hospitalized patients diagnosed with HIV infection;
* Sign the informed consent voluntarily.

Exclusion Criteria:

* Severe active infection requiring parenteral antibiotics or antifungal treatment within 30 days before the assessment;
* Other major chronic diseases that may affect health-related quality of life, such as extrahepatic malignant tumors;
* Psychotic patients, patients with severe cognitive or neurological deficits;
* Women during pregnancy and lactation;
* Those who refuse to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PLWH crowd in Zhejiang Province
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-05-26 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of liver disease in PLWH | 2020-12-31
  The overall prevalence of liver disease in PLWH and the prevalence of hepatitis B, C, and fatty liver

CONTACTS AND LOCATIONS:
Locations (1):
- the first affiliated hospital of Zhejiang university school of medicine, Hangzhou, Zhejiang, China